CLINICAL TRIAL: NCT00172445
Title: Clinical Studies of Kikuchi's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 9361700760
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2004-06

CONDITIONS: Lymphadenitis
MeSH Terms: conditions — Lymphadenitis | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: blood sampling, neck lymph node biopsy

SUMMARY:
Kikuchi-Fujimoto disease is a distinctive syndrome of necrotizing lymphadenitis which was formally described in 1972 by two Japanese pathologists, Kikuchi and Fujimoto. It is a benign, self-limited disease that predominantly occurs in young women. It was more common in Asian people, especially in Japanese. The most frequent clinical presentations are fever (30~50%) and cervical lymphadenopathy, often tender in palpable. Other lymph node regions can be affected, and hepatosplenomegaly may be present. The laboratory findings include leucopenia with atypical lymphocytosis. ESR, transaminases and lactate dehydrogenase are often raised. The clinical features are easily confused with other conditions, particularly lymphoma. Therefore the diagnosis depends on the pathological findings. The typical findings are paracortical lesions consisting of patchy zones of eosinophilic fibrinoid necrosis and abundant karyorrhexis. In general, spontaneous resolution of symptoms and signs within a few months can be expected without treatment.For decades, the etiology of Kikuchi's disease has been speculated. Although the perforin and Fas pathways of cytotoxic T cells induce an abundance of apoptosis and thus induce necrotizing lesions, the trigger factor is unknown. Since the disease can precede or occur in association with a connective tissue disorder, especially SLE, the autoimmune contribution to the etiology has also been speculated. However, the clinical course of Kikuchi's disease, often sudden onset and spontaneous resolution, the frequent flu-like or upper respiratory prodrome, and the prominence of cervical lymphadenopathy, support a viral cause. Evidence for a viral cause also includes peripheral blood atypical lymphocytosis and elevated serum IFN-a or 2'-5' oligoadenylate synthetase levels. Several infectious agents have been suggested, including bacteria (e.g. Brucella, Yersinia), parasites (e.g. toxoplasmosis) and viruses (e.g. EBV, CMV, HHV6, HHV8, parvovirus B19, HTLV, HIV).The aim of this study is to collect cases of Kikuchi' disease in bureau of NHI and NTUH. We will analyze the incidence rate, age of onset, sex, season of onset and clinical course to see if there is any clustered cases, or nosocomial infection. Then we will study the etiology of Kikuchi's disease especially the infection causes by analyzing pathologic specimen and serology. We hope to find out the etiology of Kikuchi's disease and the new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Kikuchi's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LI-Chieh Wang, MD, Principal Investigator — National Taiwan University Hospital